CLINICAL TRIAL: NCT04272333
Title: A Phase 0 Study Using the CIVO® Platform to Evaluate Intratumoral Microdoses of Motolimod Singly and in Combination With Nivolumab in Patients With Head and Neck Cancer
Brief Title: Intratumoral Microdosing of Motolimod in HNSCC
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Partner Termination
Sponsor: Presage Biosciences (Industry)
Collaborators: Celgene (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PBI-CEL-01
Record Dates: First submitted 2020-02-10; First posted 2020-02-17 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: HNSCC
Keywords: precision oncology; intratumoral microdosing; microdose injection; microdosing; in vivo oncology; in vivo drug sensitivity; tumor microenvironment; multiplexed immunohistochemistry; head and neck cancer; SCCHN; pharmacodynamic biomarkers; CIVO
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — VTX-2337; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CIVO Microdose Injection of Motolimod and Nivolumab (Experimental): Patients who are scheduled for surgical biopsy or tumor resection surgery will be injected at least four hours to up to four days prior to surgery using the CIVO device. Each needle of the CIVO device will deliver up to 8.3 microliters of solution, including a vehicle control (sterile saline) or subtherapeutic microdoses of motolimod, nivolumab, or motolimod combined with nivolumab. Each microdose is simultaneously injected in a columnar fashion through each of 8, 5, or 3 needles (in a device configuration determined by tumor dimensions) into a single solid tumor or effaced metastatic lymph node.
  Interventions: Drug: Motolimod; Biological: Nivolumab; Combination Product: Motolimod + Nivolumab

INTERVENTIONS:
Drug: Motolimod — Intratumoral microdose injection by the CIVO device.
  Other Names: VTX2337
Biological: Nivolumab — Intratumoral microdose injection by the CIVO device.
  Other Names: Opdivo
Combination Product: Motolimod + Nivolumab — Intratumoral microdose injection by the CIVO device.

SUMMARY:
This is a multi-center, single arm, open-label, multi-agent, localized pharmacodynamic biomarker Phase 0 trial designed to study the biological effects within the tumor microenvironment of motolimod and motolimod combined with nivolumab when administered intratumorally in microdose quantities via the CIVO device in patients with head and neck squamous cell carcinoma (HNSCC). CIVO stands for comparative in vivo oncology.

DETAILED DESCRIPTION:
CIVO is a research tool composed of a hand-held single-use sterile injector coupled with fluorescent tracking microspheres called CIVO GLO that mark the sites of drug microdose injection, enabling rapid assessment of multiple oncology drugs or drug combinations simultaneously within a patient's tumor. In this Phase 0 intratumoral microdosing study in human patients with pathologic diagnosis of HNSCC with at least one lesion (primary, recurrent, or effaced metastatic lymph nodes) for which there is a planned surgical intervention, we will evaluate motolimod's ability to activate immune effector cells within the local tumor microenvironment. Additionally, this study will examine motolimod in combination with nivolumab to study whether motolimod enhances the localized immune responses compared to those of either immunotherapy alone. Motolimod singly and in combination with nivolumab will be delivered intratumorally in subtherapeutic microdose quantities via CIVO.

The CIVO device penetrates solid tumors and delivers subtherapeutic microdoses of up to eight anti-cancer agents or combinations of anti-cancer agents co-injected with CIVO GLO into discrete regions of the tumor. At the time of the planned surgical intervention (at least four hours to up to four days after the CIVO microdose injection), the injected tumor tissue is then excised and tumor responses are assessed via histological staining of tumor cross-sections sampled perpendicular to each injection column. Co-injection with CIVO GLO enables identification of each injection site during resection as well as in tissues stained for analysis. Because the platform delivers microdose amounts of each test agent or combination directly into the patient's tumor tissue, hypotheses can be tested earlier in the drug development process, consistent with the goals of the 2006 FDA Exploratory IND Guidance for Industry.

ELIGIBILITY:
Inclusion Criteria:

1. Ability and willingness to comply with the study's visit and assessment schedule.
2. Male or female ≥ 18 years of age at Visit 1 (Screening).
3. Pathologic diagnosis of HNSCC.
4. Ability and willingness to provide written informed consent. Voluntary written consent must be given before performance of any study related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
5. At least one lesion (primary or recurrent tumor) ≥ 2 cm in the shortest diameter that is accessible for ultrasound-guided percutaneous CIVO injection and for which there is a planned surgical intervention. An effaced metastatic lymph node may only be selected with prior Sponsor approval. Treatment plan may include adjuvant radiation or chemotherapy, and subjects should have no medical contraindication to surgery.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
7. Female patients who :

   * Are postmenopausal for at least 24 consecutive months (i.e., have not had menses at any time during the preceding 24 consecutive months), OR
   * Are surgically sterile, OR
   * Are of childbearing potential (FCBP) who agree to true abstinence from heterosexual intercourse (which must be source documented) or to use a highly effective contraceptive method (e.g., combined [containing estrogen and progestogen] or progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, intravaginal, patch, or implantable]; bilateral tubal ligation; intrauterine device; intrauterine hormone-releasing system; or vasectomized partner sterilization [note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success]) from the time of signing the Informed Consent Form (ICF) and during study participation.
   * Agree to refrain from donating ova during study participation.

Male patients who:

* Agree to practice true abstinence from heterosexual intercourse or agree to use a condom (a latex condom is recommended) during sexual contact with a pregnant female or a FCBP from the time of signing the ICF and while participating in the study, even if he has undergone a successful vasectomy.
* Agree to refrain from donating sperm during study participation.

Exclusion Criteria:

1. Tumors or effaced nodes that are anticipated by the Investigator to lack a sufficient volume of viable tumor tissue (based on available pre-operative imaging, pre-injection ultrasound imaging, or pathology reports) for CIVO injection due to size, location, necrosis, cysts, excessive stroma, fibrosis, or treatment-induced tissue changes. Lesions that have received neoadjuvant radiation therapy may lack sufficient viable tumor tissue for CIVO injection procedures.
2. Tumors near or involving critical structures for which, in the opinion of the treating clinician, injection would pose undue risk to the patient.
3. Patients with a diagnosis of nasopharyngeal carcinoma.
4. Female patients who are:

   * Both lactating and breastfeeding, OR
   * Have a positive urine β-subunit of human chorionic gonadotropin (β-hCG) pregnancy test at screening verified by the Investigator.
5. Any uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives.
6. Patients with a history of concurrent second cancers requiring active, ongoing systemic treatment.
7. Patients with active autoimmune diseases requiring treatment.
8. Patients with known human immunodeficiency virus/acquired immune deficiency syndrome (HIV/AIDS) with uncontrolled viral load and CD4 less than 200, or known chronic hepatitis B/C.
9. Patients that have received a live vaccine within 4 weeks of the baseline/screening visit.
10. Use of any of the following ≤ 2 weeks prior to CIVO injection :

    1. Chronic systemic immunosuppressive therapy or corticosteroids (e.g., prednisone or equivalent exceeding a total dose of 140 mg over the last 14 days). Intranasal, inhaled, topical, or local corticosteroid injections (e.g., intra-articular injection), or steroids as premedication for hypersensitivity reactions (e.g., computed tomography [CT] scan premedication) are exceptions to this criterion.
    2. Biological response modifiers for treatment of active autoimmune disease.
    3. Hematopoietic growth factors.
    4. Anticoagulants such as warfarin or low-molecular-weight heparin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Quantification of Cell Death and Immune Cell Biomarkers by Immunohistochemistry (IHC) and In-Situ Hybridization (ISH) in Resected Tissue | 4 hours-4 days after microdose injection
  Quantification of biomarker-positive and biomarker-negative cells will be performed within the tumor microenvironment around each of the injection sites of each resected patient sample by IHC and ISH. An aggregate analysis of this quantification may be done across patient samples to evaluate trends in tumor response. List of biomarkers evaluated may include biomarkers for cell death (e.g. cleaved caspase 3), T-cells (e.g. CD3, CD8/Granzyme B), and natural killer (NK)/myeloid cells (e.g. CD56/Granzyme B, CD86, CD68, CD163).

SECONDARY OUTCOMES:
Number of Patients with Adverse Events | Up to 28 days after microdose injection
  Relationship of AE to study drug or CIVO device will be determined using an AE Relatedness Grading System.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Presage Biosciences
Locations (5):
- United States (5):
  - University of California, San Francisco, San Francisco, California
  - University of Illinois at Chicago, Chicago, Illinois
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oregon Health & Science University (OHSU), Portland, Oregon
  - Portland VA, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klinghoffer RA, Bahrami SB, Hatton BA, Frazier JP, Moreno-Gonzalez A, Strand AD, Kerwin WS, Casalini JR, Thirstrup DJ, You S, Morris SM, Watts KL, Veiseh M, Grenley MO, Tretyak I, Dey J, Carleton M, Beirne E, Pedro KD, Ditzler SH, Girard EJ, Deckwerth TL, Bertout JA, Meleo KA, Filvaroff EH, Chopra R, Press OW, Olson JM. A technology platform to assess multiple cancer agents simultaneously within a patient's tumor. Sci Transl Med. 2015 Apr 22;7(284):284ra58. doi: 10.1126/scitranslmed.aaa7489. PMID 25904742
- [Background] Frazier JP, Bertout JA, Kerwin WS, Moreno-Gonzalez A, Casalini JR, Grenley MO, Beirne E, Watts KL, Keener A, Thirstrup DJ, Tretyak I, Ditzler SH, Tripp CD, Choy K, Gillings S, Breit MN, Meleo KA, Rizzo V, Herrera CL, Perry JA, Amaravadi RK, Olson JM, Klinghoffer RA. Multidrug Analyses in Patients Distinguish Efficacious Cancer Agents Based on Both Tumor Cell Killing and Immunomodulation. Cancer Res. 2017 Jun 1;77(11):2869-2880. doi: 10.1158/0008-5472.CAN-17-0084. Epub 2017 Mar 31. PMID 28364003
- [Background] Dey J, Kerwin WS, Grenley MO, Casalini JR, Tretyak I, Ditzler SH, Thirstrup DJ, Frazier JP, Pierce DW, Carleton M, Klinghoffer RA. A Platform for Rapid, Quantitative Assessment of Multiple Drug Combinations Simultaneously in Solid Tumors In Vivo. PLoS One. 2016 Jun 30;11(6):e0158617. doi: 10.1371/journal.pone.0158617. eCollection 2016. PMID 27359113
- [Background] Moreno-Gonzalez A, Olson JM, Klinghoffer RA. Predicting responses to chemotherapy in the context that matters - the patient. Mol Cell Oncol. 2015 Jun 10;3(1):e1057315. doi: 10.1080/23723556.2015.1057315. eCollection 2016 Jan. PMID 27308571
- [Background] Gundle KR, Deutsch GB, Goodman HJ, Pollack SM, Thompson MJ, Davis JL, Lee MY, Ramirez DC, Kerwin W, Bertout JA, Grenley MO, Sottero KHW, Beirne E, Frazier J, Dey J, Ellison M, Klinghoffer RA, Maki RG. Multiplexed Evaluation of Microdosed Antineoplastic Agents In Situ in the Tumor Microenvironment of Patients with Soft Tissue Sarcoma. Clin Cancer Res. 2020 Aug 1;26(15):3958-3968. doi: 10.1158/1078-0432.CCR-20-0614. Epub 2020 Apr 16. PMID 32299817
- See also: Presage Website — https://presagebio.com/